CLINICAL TRIAL: NCT07307430
Title: Effect of a Structured Narrative Education Program on Glycemic Control in Adults With Type 2 Diabetes in Primary Care: A Randomized Controlled Trial
Brief Title: Effect of Narrative Education on Glycemic Control in Adults With Type 2 Diabetes in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Veli BİLEN, Research Assistant, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMKU-FM-NARRATIVE-T2DM-2026
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Diabetes Self-management; Diabetes Education
Keywords: Primary care; Narrative education; Diabetes self-management; HbA1c; Randomized controlled trial; Self-care behaviors; SDSCA; PAID-5; Family medicine; Behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group design with 1:1 assignment to standard care versus structured narrative education plus standard care.
Masking Description: Due to the nature of the intervention, participants and care providers are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants receive usual diabetes care and routine counseling in primary care; no structured narrative education sessions are provided.
- Narrative Education + Standard Care (Experimental): Participants receive usual care plus a structured narrative education program over 3 months (two individual face-to-face sessions at Day 0 and Day 15 and four brief reinforcement phone calls at Days 30, 45, 60, and 75).
  Interventions: Behavioral: Structured Narrative Education Program

INTERVENTIONS:
Behavioral: Structured Narrative Education Program — Two individual face-to-face narrative sessions (20-30 minutes) at Day 0 and Day 15 plus four brief reinforcement phone calls (3-5 minutes) at Days 30, 45, 60, and 75 to support diabetes self-care goal setting and adherence.
  Other Names: Narrative Education
  Arms: Narrative Education + Standard Care

SUMMARY:
Type 2 diabetes is common in primary care, and daily self-care behaviors are essential for achieving blood sugar targets. This randomized, two-arm clinical trial will evaluate whether a structured narrative education program added to usual diabetes care improves glycemic control compared with usual care alone in adults with type 2 diabetes. Eligible participants (age ≥18 years) with suboptimal glycemic control (HbA1c ≥7.0% in the last 3 months) will be randomized 1:1 to either standard care or standard care plus narrative education. The narrative education program will be delivered by a family physician over 3 months and includes two individual face-to-face sessions (approximately 20-30 minutes) at Day 0 and Day 15 and four brief telephone reinforcement calls (approximately 3-5 minutes) on Days 30, 45, 60, and 75.

The primary outcome is the absolute change in HbA1c from baseline (Day 0) to Day 90. Secondary outcomes include changes in diabetes self-care activities (SDSCA-TR), diabetes-related distress (PAID-5-TR), and body mass index (BMI) from Day 0 to Day 90.

DETAILED DESCRIPTION:
This single-center, parallel-group randomized controlled trial will be conducted in a primary care family health center. After eligibility assessment and written informed consent, participants will be randomized 1:1 to the Narrative Education Group (intervention) or the Standard Care Group (control). Randomization will be generated by an independent third person not involved in the conduct of the study using computer-based block randomization (block size 4 or 6). Allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes opened in the presence of the participant after consent. Because of the nature of the intervention, participants and the clinician delivering the sessions cannot be blinded; however, data entry and statistical analyses will be performed using coded groups.

Both groups will continue to receive routine diabetes management provided by the family physician and/or relevant specialists; the study protocol will not dictate medication initiation or changes. The control group will not receive any additional structured education sessions beyond routine counseling.

Participants in the intervention group will receive a structured narrative education program over approximately 3 months, consisting of two individual face-to-face sessions (about 20-30 minutes) at Day 0 and Day 15 and four brief telephone reinforcement calls (about 3-5 minutes) at Days 30, 45, 60, and 75. Face-to-face sessions emphasize the patient's personal experience of living with diabetes using open-ended reflective questions, with the goal of increasing awareness, identifying barriers, and setting small, achievable behavior goals. Telephone calls are used for reinforcement and appointment reminders; no measurements or questionnaires are administered during these calls.

Assessments will be performed at baseline (Day 0) and at 3 months (Day 90). At both time points, HbA1c and BMI will be recorded, and the SDSCA-TR and PAID-5-TR questionnaires will be administered. The primary outcome is the absolute change in HbA1c from Day 0 to Day 90. Secondary outcomes are changes in SDSCA-TR, PAID-5-TR, and BMI from Day 0 to Day 90. Process indicators (e.g., adherence to planned sessions and Day 90 follow-up rate) will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of type 2 diabetes mellitus for at least 1 year
* HbA1c ≥ 7.0% measured within the last 3 months prior to enrollment
* Followed in the study family health center and reachable by telephone
* Able to read and write (or able to complete questionnaires with investigator assistance)
* Provides written informed consent

Exclusion Criteria:

* Type 1 diabetes, gestational diabetes, or secondary diabetes
* Acute infection or hospitalization within the last 2 weeks
* Major surgery or blood transfusion within the last 3 months
* Active malignancy or current systemic steroid/immunosuppressive therapy
* Significant cognitive impairment preventing participation
* Current participation in another structured diabetes education program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (%) | Baseline (Day 0) to Day 90
  Absolute change in glycated hemoglobin (HbA1c) from baseline (Day 0) to Day 90.

SECONDARY OUTCOMES:
Change in Summary of Diabetes Self-Care Activities (SDSCA) total score | Baseline (Day 0) to Day 90
  Summary of Diabetes Self-Care Activities (SDSCA), Turkish version (SDSCA-TR). The SDSCA is a self-report measure of diabetes self-care over the past 7 days. Total score range: 0 to 7, with higher scores indicating better self-care. The outcome is the change in SDSCA-TR total score from baseline (Day 0) to Day 90.
Change in Problem Areas in Diabetes (PAID-5) total score | Baseline (Day 0) to Day 90
  Problem Areas in Diabetes - 5 item short form (PAID-5), Turkish version (PAID-5-TR). The PAID-5 assesses diabetes-related emotional distress. Total score range: 0 to 20, with higher scores indicating greater (worse) diabetes distress. The outcome is the change in PAID-5-TR total score from baseline (Day 0) to Day 90.
Change in Body Mass Index (BMI), kg/m² | Baseline (Day 0) to Day 90
  Change in body mass index (BMI) calculated as weight (kg) / height (m²) from baseline (Day 0) to Day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Cahit ÖZER, MD, Principal Investigator — Mustafa Kemal University
Locations (1):
- Ozerli Family Health Center No. 4, Antakya, Hatay, Turkey (Türkiye)